CLINICAL TRIAL: NCT05907174
Title: Evaluating the Role of Peers to Reduce Substance Use Stigma and Improve HIV Care Outcomes in South Africa
Brief Title: Siyakhana Peer: Evaluating a Peer Recovery Coach Model to Reduce Substance Use Stigma in South African HIV Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: Medical Research Council, South Africa (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jessica Magidson, Associate Professor, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EC016-7/2022; R21DA053212 (NIH)
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Substance-Related Disorders; Substance Use; Substance Use Disorders; Stigma, Social; Stigmatization; Attitude of Health Personnel; Treatment Adherence; Treatment Adherence and Compliance; Health Care Seeking Behavior; HIV; Mental Health Recovery; Delivery of Health Care; Global Health; South Africa; Health Personnel Attitude; Health Personnel; Community Health Workers; Substance Use Recovery
Keywords: Substance-Related Disorders; Substance Use; Substance Use Disorders; Social Stigma; Substance Use Stigma; Attitude of Health Personnel; Treatment Adherence and Compliance; Health Care Seeking Behavior; HIV; Mental Health Recovery; Substance Use Recovery; Global Health; South Africa; Health Personnel; Community Health Workers
MeSH Terms: conditions — Substance-Related Disorders; Social Stigma; Stereotyping; Treatment Adherence and Compliance; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: This study uses a parallel design. Two existing teams of healthcare workers will be randomized 1:1 at the team level to either have a PRC integrated onto their team or to continue their patient care as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Enhanced Treatment as Usual (Healthcare Workers) (No Intervention): Monitoring of treatment as usual (i.e., routine interactions between healthcare workers and patients). Treatment as usual will be enhanced by providing healthcare workers with a substance use psychoeducation and screening training.
- Siyakhana - P (Healthcare Workers) (Experimental): Providers working with PRC. Siyakhana - P healthcare workers will also receive a substance use psychoeducation and screening training, and a workshop for healthcare workers to get to know the PRC and learn more about the PRC role.
  Interventions: Behavioral: Siyakhana - P
- Enhanced Treatment as Usual (Patients) (No Intervention): Monitoring of treatment as usual (i.e., routine interactions between healthcare workers and patients). Treatment as usual will be enhanced by providing healthcare workers with a substance use psychoeducation and screening training.
- Siyakhana - P (Patients) (Experimental): Patients seen by the team of health care workers with an integrated PRC. Patients will have the opportunity to meet with the PRC for about 3-months after their baseline assessment. Siyakhana - P healthcare workers will also receive a substance use psychoeducation and screening training, and a workshop for healthcare workers to get to know the PRC and learn more about the PRC role.
  Interventions: Behavioral: Siyakhana - P

INTERVENTIONS:
Behavioral: Siyakhana - P — A trained peer recovery coach (PRC) will be integrated onto the healthcare worker team randomized to Siyakhana - P. The PRC on this team will work with eligible and consenting patients who are seen by members of this healthcare team.
  Other Names: Peer Recovery Coach Integrated Intervention; PRC Integration
  Arms: Siyakhana - P (Healthcare Workers); Siyakhana - P (Patients)

SUMMARY:
Alcohol and other drug use is common among people living with HIV in South Africa and is associated with worse engagement in HIV care. There is evidence that healthcare workers in this setting, including community health workers who play a central role in re-engaging patients back into HIV care, exhibit stigmatizing behaviors towards HIV patients who use substances. In general, healthcare worker stigma towards alcohol and other drug use is associated with poorer treatment of patients who use substances, and in this setting, healthcare worker stigma towards alcohol and other drug use has been associated with worse patient engagement in HIV care. In the United States, peer recovery coaches (PRCs), who are trained individuals with lived substance use recovery experience, have helped patients who use substances engage in healthcare. Theoretically, integrating a PRC onto a healthcare team also increases healthcare worker contact with a person with substance use experience, which may be associated with lower stigma. Yet, a PRC model has not yet been tested in South African HIV care. Therefore, the purpose of this study is to develop and pilot a PRC model integrated into community-based primary care teams providing HIV services in South Africa. The study aims to compare a healthcare team with a PRC to a team without a PRC. The investigators will primarily assess the implementation of this PRC model and rates of patient re-engagement in care.

DETAILED DESCRIPTION:
South Africa has the most people living with HIV in the world, many of whom use alcohol and other drugs. Alcohol and other drug use is associated with worse HIV care engagement, contributing to increased HIV-related morbidity and mortality.

Healthcare worker stigma towards alcohol and other drug use is associated with poorer treatment of patients who use substances and worse patient engagement in HIV care. There is evidence that healthcare workers in this setting, including community health workers who play a central role in re-engaging patients who are lost to follow-up from HIV care, exhibit stigmatizing behaviors towards HIV patients who use substances.

Peer recovery coaches (PRCs) are trained individuals with lived substance use recovery experience who are integrated into healthcare teams. Healthcare workers who work with PRCs have sustained contact with a person with lived substance use experience, which is associated with lower stigma. In the United States, preliminary research has demonstrated that PRCs can be successfully integrated into healthcare teams, and that PRC contact is associated with increased patient engagement in healthcare. Yet, a PRC model has not yet been tested in South African HIV care.

Therefore, the purpose of this study is to examine the preliminary implementation and effectiveness of integrating a PRC model into existing teams of healthcare workers who are tasked with re-engaging patients in HIV care through community-based primary care teams. In a type 1, hybrid effectiveness-implementation trial, and comparing a healthcare worker team that works with a PRC to one that does not, the investigators will primarily assess the rate of patient re-engagement in care and implementation (i.e., feasibility, acceptability) of the model. Healthcare worker stigma towards patients living with HIV who use substances will also be measured.

ELIGIBILITY:
1. HEALTHCARE WORKER:

   1. Inclusion Criteria:

      * At least 18 years old
      * Employed as a healthcare worker (e.g., community health worker, nurse, supervisor, etc.,) for one of the partner healthcare worker teams that provides HIV re-engagement services
   2. Exclusion Criteria:

      * Unable or unwilling to complete informed consent and study procedures in English, isiXhosa, or Afrikaans
2. PATIENT:

   1. Inclusion Criteria:

      * At least 18 years old
      * Living with HIV
      * Problematic alcohol or other drug use defined by either: a) AUDIT-C score ≥ 2; or b) self-report illicit drug use within past 3 months
      * Seen by a healthcare worker from one of the healthcare teams partnered with this study because of recent disengagement in HIV care
   2. Exclusion Criteria:

      * Unable or unwilling to complete informed consent and study procedures in English, isiXhosa, or Afrikaans

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica F Magidson, PhD, Principal Investigator — University of Maryland, College Park; Bronwyn Myers, PhD, Principal Investigator — Medical Research Council, South Africa
Locations (1):
- South African Medical Research Council - Delft Office, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
After all primary analyses are complete, de-identified data will be available per request of outside individual
Supporting Information: Study Protocol, ICF

RESULTS

PARTICIPANT FLOW:
Period: Baseline & COPC Team-Level Randomization
Arm/Group | Enhanced Treatment as Usual (Healthcare Workers) | Siyakhana - P (Healthcare Workers) | Enhanced Treatment as Usual (Patients) | Siyakhana - P (Patients)
Started | 20 | 21 | 25 | 25
Completed | 20 | 21 | 25 | 25
Not Completed | 0 | 0 | 0 | 0
Period: 3-Month Assessment
Arm/Group | Enhanced Treatment as Usual (Healthcare Workers) | Siyakhana - P (Healthcare Workers) | Enhanced Treatment as Usual (Patients) | Siyakhana - P (Patients)
Started | 20 | 21 | 25 | 25
Completed | 19 (n=1 pt was on leave from work during assessment a study team was unable to contact for assessment. Considered Lost to Follow-up for this assessment only. Pt was still eligible for next assessment.) | 20 (n=1 pt changed jobs and study team was unable to contact for assessment. Considered Lost to Follow-up for this assessment only. Pt was still eligible for subsequent assessments.) | 24 (n=1: study team unable to contact pt for assessment. Considered Lost to Follow-up for this assessment only. Pt was still eligible for next assessment.) | 23 (n=1: study team unable to contact pt for assessment. Considered Lost to Follow-up for this assessment only. Pt was still eligible for next assessment. n=1 pt told study team they no longer wanted to participate in study. Pt considered Withdrawn by Subject and not eligible for next assessment.)
Not Completed | 1 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1
Period: 6-Month Assessment
Arm/Group | Enhanced Treatment as Usual (Healthcare Workers) | Siyakhana - P (Healthcare Workers) | Enhanced Treatment as Usual (Patients) | Siyakhana - P (Patients)
Started | 20 (Participants eligible for this assessment even if they missed the previous assessment.) | 21 (Participants eligible for this assessment even if they missed the previous assessment.) | 25 (Participants eligible for this assessment even if they missed the previous assessment.) | 24 (Participants eligible for this assessment even if they missed the previous assessment. n=1 participant withdrew from study, and therefore, was not considered eligible for this assessment.)
Completed | 20 | 20 (n=1 pt changed jobs and study team was unable to contact for assessment.) | 20 (n=3 pts passed away between their previous assessment and this assessment (non-study related) n=1 pt moved to a different province and study team was unable to contact for assessment. Considered Lost to Follow-Up. n=1 pt told study team they no longer wanted to participate in study. Considered Withdrawn by Subject.) | 22 (n=1: study team unable to contact pt for assessment. Considered Lost to Follow-Up. n=1 pt told study team they no longer wanted to participate in study. Pt considered Withdrawn by Subject.)
Not Completed | 0 | 1 | 5 | 2
Not completed — Death | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Treatment as Usual (Healthcare Workers) | Siyakhana - P (Healthcare Workers) | Enhanced Treatment as Usual (Patients) | Siyakhana - P (Patients) | Total
Number analyzed (Participants) | 20 | 21 | 25 | 25 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.10 (9.75) | 43.33 (8.59) | 44.88 (8.53) | 41.84 (10.91) | 42.86 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 24 | 19 | 83
  Male | 0 | 1 | 1 | 6 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black African | 20 | 18 | 23 | 21 | 82
  Race: Coloured (South African category) | 0 | 3 | 2 | 4 | 9
Region of Enrollment [Number; unit: participants]
  South Africa | 20 | 21 | 25 | 25 | 91

OUTCOME MEASURES:

1. Primary Outcome: Healthcare Worker Substance Use Stigma
Description: Healthcare worker stigma towards substance use measured using the Social Distance Scale (SDS). SDS scores range from 6 to 24, with higher scores indicating more desired social distance (higher stigma).
Time Frame: 3-months post-baseline assessment
Population: Only healthcare worker participants completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Treatment as Usual (Healthcare Workers) | Siyakhana - P (Healthcare Workers) | Enhanced Treatment as Usual (Patients) | Siyakhana - P (Patients)
Number analyzed (Participants) | 19 | 20 | 0 | 0
score on a scale | 11.63 (2.87) | 9.95 (2.93) |  |
Statistical Analysis 1: Comparison: Enhanced Treatment as Usual (Healthcare Workers) vs Siyakhana - P (Healthcare Workers); Test type: Superiority; p = 0.023, Regression, Linear; B = -2.23

2. Secondary Outcome: Healthcare Worker Feasibility (Intervention Arm Only)
Description: Feasibility subscale of the JHU Applied Mental Health Research (AMHR) D&I Measure, a 10-item measure for assessing dissemination and implementation outcomes in low- and middle-income settings, completed by healthcare worker participants. Items are rated on a 0-3 scale, and averaged, with lower scores (closer to 0) indicating lower feasibility and higher scores (closer to 3) indicating higher feasibility. Findings will be supplemented with qualitative interviews.
Time Frame: 6-months post-integration assessment
Population: Only healthcare participants in the Siyakhana-P condition completed this measure. Of the n = 20 who completed the 6-month assessment, n = 2 never worked directly with the PRC and therefore did not complete this measure. Therefore, data from n = 18 participants was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Treatment as Usual (Healthcare Workers) | Siyakhana - P (Healthcare Workers) | Enhanced Treatment as Usual (Patients) | Siyakhana - P (Patients)
Number analyzed (Participants) | 0 | 18 | 0 | 0
score on a scale |  | 2.35 (0.63) |  |

3. Secondary Outcome: Healthcare Worker Acceptability (Intervention Arm Only)
Description: Acceptability subscale of the JHU Applied Mental Health Research (AMHR) D&I Measure, a 14-item measure for assessing dissemination and implementation outcomes in low- and middle-income settings, completed by healthcare worker participants. Items are rated on a 0-3 scale, and averaged, with lower scores (closer to 0) indicating lower acceptability and higher scores (closer to 3) indicating higher acceptability. Findings will be supplemented with qualitative interviews.
Time Frame: 6-months post-integration assessment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Treatment as Usual (Healthcare Workers) | Siyakhana - P (Healthcare Workers) | Enhanced Treatment as Usual (Patients) | Siyakhana - P (Patients)
Number analyzed (Participants) | 0 | 18 | 0 | 0
score on a scale |  | 2.46 (0.58) |  |

4. Other Pre Specified Outcome: Patient Re-Engagement in HIV Care
Description: Patient HIV care re-engagement (dichotomous yes/no), assessed via clinic records.
Time Frame: 3-months post-baseline assessment
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Patient Feasibility (Intervention Arm Only)
Description: Feasibility subscale of the JHU Applied Mental Health Research (AMHR) D&I Measure, a 14-item measure for assessing dissemination and implementation outcomes in low- and middle-income settings, completed by patient participants. Items are rated on a 0-3 scale, and averaged, with lower scores (closer to 0) indicating lower feasibility and higher scores (closer to 3) indicating higher feasibility. Findings will be supplemented with qualitative interviews.
Time Frame: 3-months post-baseline assessment
Population: Only patient participants in the Siyakhana - P intervention condition completed this measure. Of the n=23 Siyakhana - P patient participants who completed the 3-Month Assessment, n=1 never met with the PRC and therefore did not answer the questions. Therefore, a total of n=22 participants are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Treatment as Usual (Healthcare Workers) | Siyakhana - P (Healthcare Workers) | Enhanced Treatment as Usual (Patients) | Siyakhana - P (Patients)
Number analyzed (Participants) | 0 | 0 | 0 | 22
score on a scale |  |  |  | 2.77 (0.24)

6. Other Pre Specified Outcome: Patient Acceptability (Intervention Arm Only)
Description: Acceptability subscale of the JHU Applied Mental Health Research (AMHR) D&I Measure, a 12-item measure for assessing dissemination and implementation outcomes in low- and middle-income settings, completed by patient participants. Items are rated on a 0-3 scale, and averaged, with lower scores (closer to 0) indicating lower acceptability and higher scores (closer to 3) indicating higher acceptability. Findings will be supplemented with qualitative interviews.
Time Frame: 3-months post-baseline assessment
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Treatment as Usual (Healthcare Workers) | Siyakhana - P (Healthcare Workers) | Enhanced Treatment as Usual (Patients) | Siyakhana - P (Patients)
Number analyzed (Participants) | 0 | 0 | 0 | 22
score on a scale |  |  |  | 2.86 (0.28)

ADVERSE EVENTS:
Time Frame: Adverse events are monitored an average of 15 months for each participant, from signing of informed consent to the final follow-up.
Arm/Group | Enhanced Treatment as Usual (Healthcare Workers) | Siyakhana - P (Healthcare Workers) | Enhanced Treatment as Usual (Patients) | Siyakhana - P (Patients)
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/21 | 3/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/21 | 4/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/25 | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Treatment as Usual (Healthcare Workers) (N=20) | Siyakhana - P (Healthcare Workers) (N=21) | Enhanced Treatment as Usual (Patients) (N=25) | Siyakhana - P (Patients) (N=25)
Death (General disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) — Death, cause unknown (family/friends reported they did not know the cause of death)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — 5-day hospitalization due to pulmonary tuberculosis (diagnosed during hospital stay).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Treatment as Usual (Healthcare Workers) (N=20) | Siyakhana - P (Healthcare Workers) (N=21) | Enhanced Treatment as Usual (Patients) (N=25) | Siyakhana - P (Patients) (N=25)
Birth in hospital, infant death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pt admitted to hospital to give birth (planned). Infant did not survive. Pt discharged from hospital shortly after.
Suicidal Thoughts (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pt reported suicidal thoughts during a qualitative interview. Study staff accompanied pt to clinic to meet with a psychologist.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT05907174/Prot_SAP_000.pdf